CLINICAL TRIAL: NCT03017417
Title: A COMbined progRamme of Exercise and Dietary ADvice in mEn With Castrate Resistant Prostate Cancer - COMRADE Trial
Brief Title: A COMbined progRamme of Exercise and Dietary ADvice in mEn With Castrate Resistant Prostate Cancer
Acronym: COMRADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STH19598
Record Dates: First submitted 2016-11-14; First posted 2017-01-11 (Estimated); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Prostatic Neoplasms, Castration-Resistant; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention arm (Experimental): exercise training intervention to include:
  * DEXA scan will collect data on via a full body scan to determine post-cranial appendicular whole body LM, whole body fat free mass (FFM) and whole body FM.
  * Muscle Strength assessment
  * Physical function assessment
  * Questionnaires and diet diaries
  Interventions: Other: Exercise Intervention
- standard of care arm (Active Comparator): * standard treatment
  * exercise advice
  * Questionnaires
  Interventions: Other: standard of care

INTERVENTIONS:
Other: Exercise Intervention — Various exercise tests
  Arms: Exercise Intervention arm
Other: standard of care — standard treatment
  Arms: standard of care arm

SUMMARY:
The proposed study will assess the feasibility of an exercise and dietary intervention in men with castrate resistant prostate cancer with secondary outcomes assessing improvements in physical functioning, fatigue, quality of life, and body composition.The study will have 2 arms, with one set of participants randomized to resistance exercise training intervention plus dietary advice and the other arm will be standard of care plus exercise advice.

DETAILED DESCRIPTION:
Although there have been advances in recent years, therapeutic options remain limited for men with castrate resistant prostate cancer (CRPC). There is an unmet clinical need for interventions which can improve quality of life, functional capacity and cancer related fatigue. Adjunctive exercise therapy could be a potentially effective treatment for these men. A growing body of evidence has demonstrated numerous benefits in physiological and psychosocial outcomes in men with advanced prostate cancer. Further, there is observational evidence linking physical activity with reduced disease specific mortality after a diagnosis of cancer. Observational data also indicates that preserving skeletal muscle mass can improve responses to chemotherapy. The proposed study will assess the feasibility of an exercise and dietary intervention in men with castrate resistant prostate cancer with secondary outcomes assessing improvements in physical functioning, fatigue, quality of life, and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Men with Castrate resistant prostate cancer
* Men with histologically confirmed PCa on long-term ADT with either

  * PSA>2ng/ml above nadir or PSA level that has risen serially on at least two occasions (each at least 4 weeks apart) in the presence of castrate levels of testosterone or;
  * Evidence of symptomatic disease progression whilst undergoing first line androgen deprivation therapy (ADT) in the presence of castrate levels of testosterone or;
  * Radiographic disease progression whilst undergoing first line ADT in the presence of castrate levels of testosterone

Exclusion Criteria:

* • Participation in other trials which might bias the evaluation of the primary objectives of the present study.

  * Current participation in regular physical activity (defined as purposeful physical activity of a moderate intensity for 90 minutes per week for at least six months).
  * Unstable angina, uncontrolled hypertension, recent myocardial infarction, pacemakers.
  * Uncontrolled painful or unstable bony metastatic lesions.
  * Within two months of invasive surgical treatment (transurethral surgery allowed).
  * Any physical, neurological or psychiatric impairment or disease or other condition that would limit the ability to understand and complete the study assessments and complete the required questionnaires, recall and record of dietary information would be excluded.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited who complete the intervention | 16 Weeks

SECONDARY OUTCOMES:
Number of participants who show improvement in the Physical function assessments | 16 weeks
number of participants who show improvement from treatment as shown by a DEXA scan | 16 weeks
number of participants who show an increase in Muscle hypertrophy following intervention assessment | 16 weeks
number of participants who show increases in Muscle Strength following intervention assessment | 16 weeks
number of participants who show a higher score on Quality of life assessments following intervention | 16 weeks
number of participants who adhere to the Diet diaries | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share data